CLINICAL TRIAL: NCT04663971
Title: IBD Audit on Fertility, Pregnancy and Delivery in Patients With Inflammatory Bowel Disease: a International Study
Brief Title: Fertility and Pregnancy After Surgery IBD Audit
Acronym: Fertile-IBD
Status: Recruiting | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: University of Bologna (Other); University of Rome Tor Vergata (Other); Italian Group for the study of Inflammatory Bowel Disease (IG-IBD) (Other)
Responsible Party: Principal Investigator, Gianluca Pellino, Lecturer, University of Campania Luigi Vanvitelli
Other Study IDs: Fertile-IBD
Record Dates: First submitted 2020-11-27; First posted 2020-12-11 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Fertility Disorders; Pregnancy Complications; Delivery Problem
Keywords: Crohn's disease; ulcerative colitis; surgery
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Pregnancy Complications; Dystocia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crohn's disease: Patients with Crohn's disease.
  Interventions: Procedure: Any surgery; Procedure: Any medical treatment
- Ulcerative colitis: Patients with Ulcerative colitis
  Interventions: Procedure: Any surgery; Procedure: Any medical treatment

INTERVENTIONS:
Procedure: Any surgery — Any surgical procedures performed for inflammatory bowel diseases
Procedure: Any medical treatment — Any treatment (including non-surgical) performed for inflammatory bowel diseases

SUMMARY:
Crohn's disease and Ulcerative colitis are chronic disease that are usually diagnosed at young age. The diseases and the associated treatment can impact on patient's sexual function, fertility, pregnancy, and delivery. This study aims to assess the impact of inflammatory bowel diseases on these aspects in female patients.

DETAILED DESCRIPTION:
This is a cross-sectional, international, multicentre study. Female patients diagnosed with inflammatory bowel diseases (Crohn's disease and ulcerative colitis) treated at several Italian centres will be retrospectively assessed for inclusion.

Those who underwent surgery below the age of 35 years between 2000 and 2020 will be included. The study aims to obtain information on female fertility, pregnancy and delivery, and to identify factors associated with infertility and problems to conclude the pregnancy.

For each nation, at least one centre will collect data on patients who were not treated with surgery.

Patients who meet inclusion criteria will be asked to prospectively fill a questionnaire on fertility and pregnancy.

Data on treatments and demographic will be retrospectively collected by the local investigators and uploaded on a secure online database.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease diagnosis
* ulcerative disease diagnosis
* operated on before 36 years of age

Exclusion Criteria:

* younger than 18 years old at follow-up
* no definitive diagnosis
* no surgical procedures performed

A subgroup of patients who did not undergo surgery will be used, at least one for each country.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All female patients will be included
Study Population: Female patients diagnosed with Crohn's disease or ulcerative colitis, treated when 35-year-old or younger.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Fertility | through study completion, an average of 1 year
  Rate of infertility and number of pregnancies. Number of attempts to achieve pregnancy.
Pregnancy | through study completion, an average of 1 year
  Rate of successful pregnancies. Number of miscarriages.

SECONDARY OUTCOMES:
In-vitro fertilization | through study completion, an average of 1 year
  Number of in-vitro fertilization attempts
Abortion/s | through study completion, an average of 1 year
  Number of abortions and reasons.
Complications, surgical | through study completion, an average of 1 year
  Incidence of early and late surgical complications and effects on fertility
Complications, medical | through study completion, an average of 1 year
  Incidence of medical complications and effects on fertility
Surgical approach | through study completion, an average of 1 year
  Rate of minimally invasive surgery use and effect on fertility and pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Sica, MD, PhD, Study Chair — University Tor Vergata Roma; Matteo Rottoli, MD, PhD, Study Chair — University Alma Mater Bologna; Francesco Selvaggi, MD, PhD, Study Chair — University of Campania Luigi Vanvitelli Napoli
Locations (4):
- Italy (4):
  - Policlinico S.Orsola-Malpighi, Bologna
  - Rho Memorial Hospital, Milan
  - Universitá degli Studi della Campania Luigi Vanvitelli, Napoli
  - Policlinico Tor Vergata, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] M Rottoli, P Pezzuto, G Fallani, G Pellino, F Rizzello, P Gionchetti, G Poggioli. P199 Ileal pouch-anal anastomosis in women of childbearing age affected by ulcerative colitis: a single-centre study on the risk factors for infertility and outcomes of pregnancy over 17 years. Journal of Crohn's and Colitis, Volume 16, Issue Supplement_1, January 2022, Pages i259-i261, https://doi.org/10.1093/ecco-jcc/jjab232.326
- [Result] Bernell O, Lapidus A, Hellers G. Risk factors for surgery and recurrence in 907 patients with primary ileocaecal Crohn's disease. Br J Surg. 2000 Dec;87(12):1697-701. doi: 10.1046/j.1365-2168.2000.01589.x. PMID 11122187
- [Result] Spinelli A, Sacchi M, Bazzi P, Leone N, Danese S, Montorsi M. Laparoscopic surgery for recurrent Crohn's disease. Gastroenterol Res Pract. 2012;2012:381017. doi: 10.1155/2012/381017. Epub 2012 Jan 2. PMID 22253619
- [Result] Cosnes J, de Parades V, Carbonnel F, Beaugerie L, Ngo Y, Gendre JP, Sezeur A, Gallot D, Malafosse M, le Quintrec Y. Classification of the sequelae of bowel resection for Crohn's disease. Br J Surg. 1994 Nov;81(11):1627-31. doi: 10.1002/bjs.1800811122. PMID 7827890
- [Result] Pellino G, Keller DS, Sampietro GM, Carvello M, Celentano V, Coco C, Colombo F, Geccherle A, Luglio G, Rottoli M, Scarpa M, Sciaudone G, Sica G, Sofo L, Zinicola R, Leone S, Danese S, Spinelli A, Delaini G, Selvaggi F; Italian Society of Colorectal Surgery SICCR. Inflammatory bowel disease position statement of the Italian Society of Colorectal Surgery (SICCR): ulcerative colitis. Tech Coloproctol. 2020 May;24(5):397-419. doi: 10.1007/s10151-020-02175-z. Epub 2020 Mar 2. PMID 32124113
- [Result] Calvet X, Panes J, Alfaro N, Hinojosa J, Sicilia B, Gallego M, Perez I, Lazaro y de Mercado P, Gomollon F; Members of Consensus Group; Aldeguera X, Alos R, Andreu M, Barreiro M, Bermejo F, Casis B, Domenech E, Espin E, Esteve M, Garcia-Sanchez V, Lopez-Sanroman A, Martinez-Montiel P, Luis Mendoza J, Gisbert JP, Vera M, Dosal A, Sanchez E, Marin L, Sanroman L, Pinilla P, Murciano F, Torrejon A, Ramon Garcia J, Ortega M, Roldan J. Delphi consensus statement: Quality Indicators for Inflammatory Bowel Disease Comprehensive Care Units. J Crohns Colitis. 2014 Mar;8(3):240-51. doi: 10.1016/j.crohns.2013.10.010. Epub 2013 Dec 2. PMID 24295646
- [Result] Rajaratnam SG, Eglinton TW, Hider P, Fearnhead NS. Impact of ileal pouch-anal anastomosis on female fertility: meta-analysis and systematic review. Int J Colorectal Dis. 2011 Nov;26(11):1365-74. doi: 10.1007/s00384-011-1274-9. Epub 2011 Jul 16. PMID 21766164
- [Result] Waljee A, Waljee J, Morris AM, Higgins PD. Threefold increased risk of infertility: a meta-analysis of infertility after ileal pouch anal anastomosis in ulcerative colitis. Gut. 2006 Nov;55(11):1575-80. doi: 10.1136/gut.2005.090316. Epub 2006 Jun 13. PMID 16772310
- [Result] Beyer-Berjot L, Maggiori L, Birnbaum D, Lefevre JH, Berdah S, Panis Y. A total laparoscopic approach reduces the infertility rate after ileal pouch-anal anastomosis: a 2-center study. Ann Surg. 2013 Aug;258(2):275-82. doi: 10.1097/SLA.0b013e3182813741. PMID 23360923
- [Result] Gorgun E, Cengiz TB, Aytac E, Aiello A, da Silva G, Goldberg JM, Holubar SD, Stocchi L, Wexner SD, Steele SR, Hull TL. Does laparoscopic ileal pouch-anal anastomosis reduce infertility compared with open approach? Surgery. 2019 Oct;166(4):670-677. doi: 10.1016/j.surg.2019.04.045. Epub 2019 Aug 14. PMID 31420214